CLINICAL TRIAL: NCT04003558
Title: Deep Learning Algorithms for Prediction of Lymph Node Metastasis and Prognosis in Breast Cancer MRI Radiomics (RBC-01)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other); Tungwah Hospital of Sun Yat-Sen University (Unknown); Southern Medical University, China (Other); Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Herui Yao, Principal Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSEC-KY-KS-2019-054-001
Record Dates: First submitted 2019-06-26; First posted 2019-07-01 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Breast Neoplasm Female; Early-stage Breast Cancer; Radiomics; Axillary Lymph Node; Survival, Prosthesis
Keywords: Early-stage Breast Cancer; Radiomics; Axillary lymph node metastasis; Tumor microenvironment; Survival; Deep learning
MeSH Terms: conditions — Breast Neoplasms; Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Sun Yat-Sen Memorial Hospital of Sun Yat-sen University: The cohort of Sun Yat-Sen Memorial Hospital of Sun Yat-sen University is a training cohort.
  Interventions: Other: No interventions
- Sun Yat-sen University Cancer Center: The cohort of Sun Yat-sen University Cancer Center is a validation cohort.
  Interventions: Other: No interventions
- Tungwah Hospital of Sun Yat-Sen University: The cohort of Tungwah Hospital of Sun Yat-Sen University is a validation cohort.
  Interventions: Other: No interventions
- Shunde hospital of southern medical university: The cohort of Shunde hospital of southern medical university is a validation cohort.
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — As this is a patient registry, there are no interventions.

SUMMARY:
This bi-directional, multicentre study aims to assess multiparametric MRI Radiomics-based prediction model for identifying metastasis lymph nodes and prognostic prediction in breast cancer.

DETAILED DESCRIPTION:
Sensitivity for prediction of lymph node metastasis and survival of currently available prognostic scores in limited. This study proposes to establish a deep learning algorithms of multiparametric MRI radiomics and nomogram for identifying lymph node metastasis and prognostic prediction of breast cancer. The study will investigate the relationship between the radiomics and the tumor microenvironment. The study includes the construction of multiparametric MRI radiomics-based prediction model and the validation of the prediction model.

ELIGIBILITY:
Inclusion Criteria:

* The primary lesion was diagnosed as invasive breast cancer
* Patients can have regional lymph node metastasis,but no distant organ metastasis
* Complete the breast MRI examination before treatment
* Accept breast cancer surgery or lymph node biopsy
* Eastern Cooperative Oncology Group performance status 0-2

Exclusion Criteria:

* Inflammatory breast cancer
* Accompanied with other primary malignant tumors
* Perform surgery,radiotherapy and lymph node biopsy before breast MRI examination
* Patients who have neoadjuvant chemotherapy
* Patients had distant and contralateral axillary lymph node metastasis
* The pathologic diagnosis was extensive ductal carcinoma in situ

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients who had early stage breast cancer and completed the breast MRI examination before operation,lymph node biopsy,neoadjuvant chemotherapy,and radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | 5 years
  Disease free survival (DFS), which defined as the time from the diagnosis of breast cancer to the confirmed time of metastatic disease, or death due to any other cause.

SECONDARY OUTCOMES:
The correlation of radiomics features and tumor microenvironment | baseline (Completed MRI data before biopsy,surgery,neoadjuvant and radiotherapy.)
  Radiomics is a tool to analyze tumor microenvironment characteristics based on breast MRI images.
Lymph node metastasis | Baseline
  The value of Radiomics of multiparametric MRI in predicting axillary lymph node metastasis.
Overall survival (OS) | 5 years
  The association between Radiomics of multiparametric MRI and overall survival (OS), which defined as the time from the beginning of diagnosis of breast cancer to the death with any causes.
Beast cancer specific motality (BCSM) | 5 years
  Defined as time between randomization and the time of death occur specific due to breast cancer
Recurrence free survival (RFS) | 5 years
  defined as time between randomization and the time of any recurrence of ipsilateral chest, breast, regional lymph node recurrence, distant metastases, or death occurred

CONTACTS AND LOCATIONS:
Overall Officials: Herui Yao, PhD, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Chuanmiao Xie, PhD, Principal Investigator — Sun Yat-sen University; Jie Ouyang, PhD, Principal Investigator — Tungwah Hospital of Sun Yat-Sen University; Qiugen Hu, PhD, Principal Investigator — Southern Medical University, China; Haotian Lin, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (5):
- China (5):
  - Tungwah Hospital of Sun Yat-Sen University, Dongguan, Guangdong
  - Shunde hospital of southern medical university, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No
Requests for the individual data or study documents will be considered where the proposed use aligns with public good purposes, does not conflict with other requests, and the requestor is willing to sign a data access agreement. Contact is though the corresponding author.

REFERENCES:
- [Derived] Yu Y, He Z, Ouyang J, Tan Y, Chen Y, Gu Y, Mao L, Ren W, Wang J, Lin L, Wu Z, Liu J, Ou Q, Hu Q, Li A, Chen K, Li C, Lu N, Li X, Su F, Liu Q, Xie C, Yao H. Magnetic resonance imaging radiomics predicts preoperative axillary lymph node metastasis to support surgical decisions and is associated with tumor microenvironment in invasive breast cancer: A machine learning, multicenter study. EBioMedicine. 2021 Jul;69:103460. doi: 10.1016/j.ebiom.2021.103460. Epub 2021 Jul 4. PMID 34233259